CLINICAL TRIAL: NCT05725486
Title: Effects of N-3 Polyunsaturated Fatty Acids Enriched Chicken Meet on Cardiovascular Function
Brief Title: N-3 Polyunsaturated Fatty Acids Enriched Chicken Meet and Cardiovascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Drenjancevic, Vice Dean for Science, Faculty of Medicine Josip Juraj Strossmayer University of Osijek, Josip Juraj Strossmayer University of Osijek
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2158614622108
Record Dates: First submitted 2023-01-24; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: n-3 Polyunsaturated Fatty Acids
Keywords: n-3 polyunsaturated fatty acids; vascular function; endothelium; oxidative stress; inflammation; microcircularion; macrocirculation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n-3 PUFA (Experimental): Intake of n-3 PUFAs enriched chicken meet for three weeks
  Interventions: Dietary Supplement: N-3 PUFAs Chicken Meet
- Control (Experimental): Intake of regular chicken meet for three weeks
  Interventions: Dietary Supplement: Regular Chicken Meet

INTERVENTIONS:
Dietary Supplement: N-3 PUFAs Chicken Meet — Intake of n-3 PUFAs enriched chicken meet for three weeks.
  Arms: n-3 PUFA
Dietary Supplement: Regular Chicken Meet — Intake of regular chicken meet for three weeks.
  Arms: Control

SUMMARY:
Evidence from multiple experimental, epidemiological, and clinical studies indicate that n-3 polyunsaturated fatty acids (n-3 PUFAs) may exert their cardiovascular (CV) protective effect, at least in part, by improving vascular endothelium-dependent function. Previously, the investigators demonstrated the significant beneficiary effect of consumption of n-3 PUFA-enriched hen eggs on microvascular endothelium-dependent reactivity, even in young healthy individuals.

The hypothesis of this research is that the consumption of n-3 PUFAs in the form of functionally enriched chicken meet has a beneficial effect on vascular reactivity measured in different vascular beds, and the lipid profile with a positive effect on the reduction of oxidative stress and inflammatory response in healthy sedentary individuals.

The main goal of this study is to investigate the influence of n-3 PUFAs functionally enriched chicken meet on vascular and endothelial function in a population of healthy young subjects and active athletes.

ELIGIBILITY:
Inclusion Criteria:

* young healthy sedentary individuals - did not perform regular physical activities for at least 12 months before conducting the study
* young healthy active athletes - have a minimum of 5 training sessions per week (mainly endurance training) for at least 12 months prior to conducting the study

Exclusion Criteria:

* smoking
* hypertension
* coronary disease
* diabetes
* hyperlipidemia
* kidney damage
* cerebrovascular and peripheral artery diseases
* and any other disease that could have an impact on vascular and endothelial function

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Microvascular endothelial function | 3 weeks
  Cutaneous microvascular blood flow will be measured by Laser Doppler Flowmetry in response to vascular occlusion (post occlusive reactive hyperaemia - PORH), in response to iontophoresis of acetylcholine (ACh) and local thermal hyperemia (LTH).
Macrovascular endothelial function | 3 weeks
  Measurement of flow mediated dilation (FMD) of brachial artery using ultrasound.
Cerebrovascular reactivity | 3 weeks
  Measurement of cerebrovascular blood flow using transcranial color Doppler (TCD).

SECONDARY OUTCOMES:
Lipid profile | 3 weeks
  Measurement of plasma cholesterol, HDL cholesterol, LDL cholesterol and triglycerides level.
Oxidative stress status | 3 weeks
  Measurement of Thiobarbituric Acid Reactive Substances (TBARS).
Systemic hemodynamics | 3 weeks
  Non-invasive assessment of systemic hemodynamics using impedance cardiography (CardioScreen 2000) - SV Stroke Volume (mL), CO Cardiac Output (L/min) and SVRI Systemic Vascular Resistance Index (dyn.s.cm-5 m2).
Serum Pro- and Anti-Inflammatory Cytokines, Chemokines, Growth Factors and Soluble Cell Adhesion Molecules Protein Concentration | 3 weeks
  Measurement of serum protein concentration (pg/mL) of various pro- and anti-inflammatory cytokines, chemokines, growth factors and soluble cell adhesion molecules by kits and panels for multiplex protein quantitation using the Luminex 200 instrument platform.
Body composition | 3 weeks
  Body composition and body fluid status measurement by a four-terminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically derived formulas (the original manufacturer's software) will be used to calculate the estimated Fat Free Mass (FFM kg) and Fat (Fat Mass kg).
Body fluid status | 3 weeks
  Body fluid status measurement by a four-terminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically derived formulas (the original manufacturer's software) will be used to calculate the estimated Total Body Water (TBW L), Extracellular Water (ECW L), Intracellular Water (ICW L), Plasma Fluid (PF L) and Interstitial Fluid (IF L).
Oxidative stress status | 3 weeks
  Measurement of Ferric-Reducing Ability of Plasma (FRAP).
Oxidative stress status | 3 weeks
  Measurement of enzyme activity assay of glutathione peroxidase (GPx).

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Center of Excellence for Personalized Health Care, Josip Juraj Strossayer University of Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: Undecided